CLINICAL TRIAL: NCT06609629
Title: Selective Lung Recruitment in Moderate to Severe ARDS : a Pilot Study
Acronym: SRIMSA
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024-A00005-42
Record Dates: First submitted 2024-07-18; First posted 2024-09-24 (Actual); Last update posted 2024-09-24 (Actual); Status verified 2024-07

CONDITIONS: Acute Respiratory Distress Syndrom
Keywords: ARDS; Recruitment maneuvers; selective recruitment maneuvers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- interventional arm (Experimental): This is a feasibility study. One arm of 10 patients is needed
  Interventions: Procedure: Selective lung recruitment

INTERVENTIONS:
Procedure: Selective lung recruitment — A bronchial blocker with a lumen is inserted in one inferior pulmonary lobe using a fibroscope. The baloon of the blocker is expended to isolate the lobe. A second ventilator is used to apply a pressure of 45cmH2o through the lumen of the blocker. The recruiting pressure is maintained 30 to 60 second. After the procedure, the blocker is removed and the procedure is repeated in the controlateral inferior lobe.

SUMMARY:
Acute respiratory distress syndrome (ARDS) is an acute condition affecting the lung after clinical aggression ( infectious process, pancreatitis, acute inflammatory event). This condition lead to major breathlessness due to the incapacity to properly oxygenize the boby because of lung lesions. Invasive mechanical ventilation is frequently required to grant sufficient oxygenation to the body. Unfortunately, while it allows oxygenation, mechanical ventilation can cause arms to the lung because of the mechanical power it delivers to the lung and create ventilation induced lung injuries (VILI). To reduce this risk, ventilator settings have been protocolized aiming to reduce the lung volume administered to the lung. It is effective to control the VILI but oxygenation may be insufficient under those protective parameters. To correct this lack of oxygenation practicians use recruiting maneuvers when a transient increase of lung volume administered to the lung to open collapse parts of the lung. Those maneuvers can cause barotrauma and provoke pneumothorax or decrease the heart flow. This study aim to assess the feasibility of selective recruitment maneuvers to increase oxygenation while reducing the risk of recruitment maneuvers.

Briefly, a dedicated bronchial blocker is introduce in a lower part of the lung, a balloon attached to the catheter is expended isolating a part of the lung and a recruiting pressure is administered through the lumen of the catheter to selectively expend the isolated part of the lung.

After the selected recruitment maneuver, the investigators will assess the expansion of the lung with a CT-scanner.

ELIGIBILITY:
Inclusion Criteria:

* acute ARDS according Berlin definition and a PaO2/FiO2 ratio inferior to 200
* patient under sedation and muscular blockade
* postero-basal consolidation on CT or pulmonary ultrasound
* affiliated to the French social insurance system

Exclusion Criteria:

* hemodynamic instability
* pregnancy
* patient under guardianship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-09-15 (Estimated); Primary Completion 2025-09 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
comparison in lung aeration before and after the recruiting manouever | the sthe second CT will be perform between hour 4 and hour 8 after the maneuver (Hour 0).
  Differance in lung aeration wil be assess with comparison between lung aeration on a chest CT-scan before the recruiting maneuver and lung aeration on a chest CT-scan after the recruitment maneuver. The principal outcome will be the ratio of normaly aerated lung volume (%)/hyperinflated lung volume (%). The higher this ratio will be the better is the recruitment (high volume recruited and low volume hyperinflated). The level of aeration of the lung will be determined using the density level on CT-scan where lung area will be classified among 4 category according a level of hounsfield unit (non aerated :density betwen +100 et -100 Hounsfield unit ; poorly aerated: density betwen -101 et -500 Hounsfield unit; normaly aerated: density betwen -501 et -900 Hounsfield unit; hyperinflated (density betwen -901 et -1000 Hounsfield unit). Each area will be quantified using AquariusTM software.

SECONDARY OUTCOMES:
difference between lung impedance before and after selective recruitment maneuvers | measured immedialtly before the recruitment maneuver (hour 0), between hour 4 to hour 8 after the recruitiment maneuver , at hour 24 after the selective recruitment maneuver
  measure of lung impedance using an electrical impedance tomodensitometry device (pulmovista Dräger)
PaO2/FiO2 ratio | measured immedialtly before the recruitment maneuver (hour 0), between hour 4 to hour 8 after the recruitiment maneuver , at hour 24 after the selective recruitment maneuver

OTHER OUTCOMES:
Occurence of pneumothorax | the second ct-scan will be perform between hour 4 and hour 8 after the recruitment maneuver (hour O). A chest-x-ray wil be perform at hour 24.
  presence of pneumothorax on the second chest CT presence of pneumothorax on chest x-ray
occurence of cardiac arrest | from enrollment to the end of treatment (from Hour 0 to Hour 24 after the recruiting maneuver)
  occurence of cardiac arrest is defined has the need of perfoming a cardio-pulmonary resuscitation
decrease in blood pressure | from the expension of the catheter ballon at the begining of the recruitment maneuvrer to the deflation of the catheter ballon at the end of the maneuver.
  defined as a drop of 20mmHg of arterial systolic pressure
decrease in peripheral O2 saturation | from the expension of the catheter ballon at the begining of the recruitment maneuvrer to the deflation of the catheter ballon at the end of the maneuver.
  mesured with a transcutaneous saturometer.

IPD SHARING:
Plan to Share IPD: No